CLINICAL TRIAL: NCT03958331
Title: Beat!: A Randomized Controlled Clinical Trial
Brief Title: Behavioral Economics and Adherence in Teens (BEAT!)
Acronym: Beat!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-8412; R21NR017633 (NIH)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Results first posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy; Adherence, Medication
Keywords: adolescents, behavioral economics, mHealth
MeSH Terms: conditions — Epilepsy; Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is 2-arm randomized controlled clinical trial to improve adherence in adolescents with epilepsy
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Automated reminders and individualized adherence feedback reports
  Interventions: Behavioral: Automated Digital Reminders; Behavioral: Individualized Adherence Feedback Report
- Treatment Group (Experimental): Automated reminders and individualized adherence feedback reports with social norms comparisons
  Interventions: Behavioral: Automated Digital Reminders; Behavioral: Individual Adherence Feedback Report with Social Norms

INTERVENTIONS:
Behavioral: Automated Digital Reminders — Reminders from electronic monitors via texts or alarms/lights
Behavioral: Individualized Adherence Feedback Report — Feedback report on individual adherence behaviors
  Arms: Control Group
Behavioral: Individual Adherence Feedback Report with Social Norms — Feedback report on individual adherence behaviors compared to other adolescents with epilepsy
  Arms: Treatment Group

SUMMARY:
Non-adherence to antiepileptic drug therapy is a significant problem for adolescents with epilepsy and has a critical impact on health and patient-reported outcomes. Evidence-based adherence interventions are lacking in this population and are critically needed. This proposal seeks to develop and evaluate a mHealth social norms adherence intervention for adolescents with epilepsy.

DETAILED DESCRIPTION:
Non-adherence to antiepileptic drugs (AEDs) is a common problem (i.e., 58% of patients have some level of non-adherence) for youth with epilepsy, with potentially devastating consequences. Adolescents with epilepsy represent a particularly vulnerable group, given their increased independence, decreased parental supervision, higher risk for deficits in organization and memory, busy and changing schedules, low motivation, and increased susceptibility to peer influence. Existing adherence interventions in epilepsy are not designed to meet the unique challenges faced by adolescents, and there are no efficacious interventions for adolescents with epilepsy. Not surprisingly, without efficacious interventions, adherence worsens during adolescence, further increasing the risk of poor health outcomes during this developmental period. While reminder strategies (e.g., automated digital reminders) are effective for the most common adherence barriers of forgetting and busy schedules, they are likely to be ineffective in increasing motivation. Leveraging social norms comparison methods (i.e., feedback about someone else's behavior related to one's own behavior) offers an opportunity to capitalize on the increased importance of peer influence while simultaneously targeting the low motivation characteristic of adolescents. Recent data in adolescents indicates that social norms interventions have incremental value and improve health behaviors above and beyond standard feedback without peer comparisons. Consistent with the ORBIT model for behavioral intervention development, our aims are to: 1) develop a feasible, accessible, and acceptable mHealth social norms intervention for improving AED adherence in adolescents with epilepsy and 2) obtain preliminary efficacy data and effect sizes for a future clinical trial. We conducted a pilot RCT of an mHealth social norms intervention (ORBIT Phase II). Adolescents with epilepsy who demonstrate non-adherence (< 95% adherence based on PI's previous RCTs; 58% of sample) during baseline will be randomized to either 1) mHealth social norms (automated digital reminders, individualized adherence feedback, and social norms feedback) or 2) control (automated digital reminders and individualized adherence feedback). Both groups will receive active intervention for five months. Primary (i.e., electronically-monitored adherence) and secondary outcomes (i.e., seizure severity, HRQOL) will be assessed post-treatment and 3 months later, respectively. If successful, the results of this study would have a large impact on pediatric epilepsy, with the potential to change clinical practice for treating non-adherence by reducing common barriers to behavioral health care. Because minimal clinician time is required, our mHealth social norms intervention also has potential for sustainability and broad dissemination for epilepsy and other pediatric conditions

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-17
* Confirmed diagnosis of epilepsy
* Antiepileptic drug monotherapy
* Ability to read and speak English

Exclusion Criteria:

* No significant developmental delay (e.g., autism, moderate/severe developmental or intellectual disability) or comorbid medical diagnoses (e.g., diabetes)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will have psychosocial, adherence, demographic, and medical data for children with epilepsy. Deidentified data can be used for many secondary analyses. Prior to sharing, all data will be de-identified in a HIPAA-compliant fashion. Data sets will be carefully reviewed to make sure that information such as age and gender cannot be used to gather additional information that could potentially identify individual subjects. For example, only year of birth, rather than the full birth date, will be made available. All categorical demographic variables will be collapsed into categories large enough so that combinations of demographic categories for age, gender, geographic location, etc., will have 10 or more individuals in each cell. All modalities of data will be shared, including raw and aggregate data. Descriptors for all variables shared will be included to prevent misuse or confusion. Any analytical methods utilized to assess the data will be defined in shared formats.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 12 months following completion of the study
Access Criteria: PI will provide the information

REFERENCES:
- [Result] Modi AC, Patel AD, Stevens J, Smith G, Huszti H, Guilfoyle SM, Mara CA, Schmidt M, Wagner JL. The psychosocial impact of COVID-19 within the first six months of the pandemic on youth with epilepsy and their caregivers. Epilepsy Behav. 2021 Apr;117:107855. doi: 10.1016/j.yebeh.2021.107855. Epub 2021 Feb 12. PMID 33636530

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We had a run-in period, in which 64 participants were not randomized to either control or treatment groups. The primary participants in this study were adolescents and caregivers did not receive the intervention. Caregivers completed parental permission (consent) forms, demographic information related to their child and provided data for two of the secondary outcomes.
Groups:
- Not Randomized (High Adherence): This group demonstrated adherence rates of >95% and thus were not randomized to either treatment arm per protocol
Period: Overall Study
Arm/Group | Control Group | Treatment Group | Not Randomized (High Adherence)
Started | 21 | 19 | 64
Completed | 14 | 17 | 47
Not Completed | 7 | 2 | 17
Not completed — Withdrawal by Subject | 3 | 1 | 5
Not completed — Weaned from medicine | 2 | 0 | 0
Not completed — Withdrawn by study staff due to non-compliance with study procedures | 2 | 1 | 12

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: No interventions were provided to these participants as they demonstrated high adherence and were not eligible for randomization based on the run-in period.
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Not Randomized | Total
Number analyzed (Participants) | 21 | 19 | 64 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.2) | 14.9 (3.2) | 15.6 (1.4) | 15.4 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 38 | 55
  Male | 13 | 10 | 26 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 18 | 62 | 101
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 13 | 15 | 58 | 86
  More than one race | 5 | 3 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 1 | 1
Monotherapy versus Polytherapy [Count of Participants; unit: Participants]
  Monotherapy | 21 | 17 | 61 | 99
  Polytherapy | 0 | 2 | 2 | 4
  Unknown | 0 | 0 | 1 | 1
Seizure Type [Count of Participants; unit: Participants]
  Focal | 5 | 7 | 9 | 21
  Generalized | 14 | 9 | 46 | 69
  Unclassified | 2 | 3 | 8 | 13
  Unknown | 0 | 0 | 1 | 1
Seizures in the Past 3 months [Count of Participants; unit: Participants]
  No | 13 | 13 | 39 | 65
  Yes | 8 | 6 | 14 | 28
  Unknown | 0 | 0 | 11 | 11
Family Insurance [Count of Participants; unit: Participants]
  Private | 10 | 17 | 43 | 70
  Public | 9 | 2 | 18 | 29
  Public and Private | 2 | 0 | 1 | 3
  Not insured | 0 | 0 | 2 | 2
Primary Caregiver [Count of Participants; unit: Participants]
  Mother/Stepmother | 16 | 16 | 51 | 83
  Father/Stepfather | 4 | 3 | 2 | 9
  Other: Grandmother, Uncle, Aunt | 1 | 0 | 0 | 1
  Unknown | 0 | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Electronically Monitored Adherence
Description: A total mean adherence rates will be calculated based on daily adherence rates captured through the SimpleMed Pillboxes or AdhereTech bottles. Scores range from 0-100%, with higher scores representing better adherence.
Time Frame: Month 7
Population: Adherence data missing for 2 participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 19 | 19
units on a scale | 45.5 (32.0) | 50.5 (37.4)
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; Test type: Superiority; p = 0.002, ANCOVA; Model controlled for baseline adherence, resistance to peer influence, dose, active seizures, COVID timing, COVID Impact (3 items), and sex; Mean Difference (Final Values) = 10.62, 95% CI 2-sided [4 to 17.25], Standard Error of Mean 3.38; We also conducted a longitudinal mixed effects model for adherence over time, estimating a groupXtime interaction with the same covariates listed above and allowing for a non-linear effect

2. Secondary Outcome: Seizure Severity-Clinician Report
Description: The Global Assessment of Severity of Epilepsy (GASE) is a one item clinician-rated measure of seizure severity. The total score ranges from 1-7, with higher scores representing more severe epilepsy
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 13 | 15
score on a scale | 2.5 (1.3) | 2.4 (1.2)

3. Secondary Outcome: Seizure Severity-Parent Report
Description: The Seizure Severity Scale-Adapted for Children is a caregiver-reported questionnaire, which is 9-items and assess seizure severity, including intrusiveness, frequency, length, and disruptiveness of seizures. A total score is calculated, ranging from 0-3, with higher scores representing worse seizure severity.
Time Frame: Month 9
Population: The number of participants analyzed does not match the participant flow as some participants did not complete this particular measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 12 | 16
score on a scale | 0.98 (0.55) | 1.11 (0.60)

4. Secondary Outcome: PedsQL Epilepsy Module - Parent Report
Description: The PedsQL-Epilepsy Module is a 29 item measure with several subscales (Impact, Cognitive, Executive Functioning, Sleep, Mood/Behavior) will be used. Scores range from 0-100 for each subscale, with higher scores representing better quality of life.
Time Frame: Month 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 13 | 16
score on a scale
  Impact (parent) | 83.3 (15.5) | 78.8 (18.0)
  Cognitive (parent) | 63.1 (28.9) | 72.4 (19.8)
  Sleep (parent) | 60.3 (17.1) | 65.1 (22.2)
  Executive functioning (parent) | 71.2 (23.2) | 72.3 (23.9)
  Mood/Behavior (parent) | 66.5 (18.5) | 67.2 (23.2)

5. Secondary Outcome: PedsQL Epilepsy Module-Adolescent Report
Description: The PedsQL Epilepsy Module is a 29-item health-related quality of life instrument with five subscales, including Impact, Cognitive, Executive Functioning, Sleep, and Mood/Behavior). Scores range from 0-100, with higher scores representing better quality of life.
Time Frame: 9-month
Population: The flow diagram differs in sample size as one less adolescent completed this measure. Thus, the sample size is n=12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 12 | 16
score on a scale
  Impact | 80 (13.5) | 82.8 (20.7)
  Cognitive | 73.6 (19.9) | 71.6 (26.1)
  Sleep | 56.9 (20.4) | 67.7 (27.2)
  Executive Functioning | 75.7 (13.5) | 65.4 (26.7)
  Mood/Behavior | 65.4 (15.1) | 71.9 (28.2)

6. Other Pre Specified Outcome: Satisfaction-Teen Report Total Score
Description: Adolescents completed this study specific Satisfaction measure, which was 23-items. This measure assesses satisfaction with the intervention content, relevance, helpfulness, and ease of use. Assessment of perceptions of the impact of what was learned from the intervention were also assessed. Eighteen of the items used a Likert format with the following ratings: Strongly Disagree, Disagree, Agree, and Strongly Agree. A total scale was calculated for the 18 items, which ranges from 18-72, with higher scores reflecting higher satisfaction. Finally, five open-ended items assessing what was most and least helpful about the intervention, what changes adolescents want to see in the intervention, and any additional input.
Time Frame: Month 7
Population: Participant numbers are lower than the Participant Flow data as some participants did not complete this particular measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 13 | 17
score on a scale | 53.5 (9.0) | 50.8 (6.0)

ADVERSE EVENTS:
Time Frame: 9 months
Description: We collected this data through medical chart review
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 3/21 | 6/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=21) | Treatment Group (N=19)
Epilepsy monitoring unit/overnight EEG (Nervous system disorders) | 1 (1) | 4 (4) — Routine overnight EEGs or Epilepsy Monitoring Unit Stays
Chest pain (Cardiac disorders) | 1 (1) | 1 (1) — Chest pain
Ear tube removal/myringoplasty (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Ear tube removal/myringoplasty
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1) — Suicidal ideation

LIMITATIONS AND CAVEATS:
Due to COVID-19, we recruited less participants than originally anticipated for the trial (n=104 versus n=138).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT03958331/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03958331/SAP_001.pdf
  • Informed Consent Form (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03958331/ICF_002.pdf